CLINICAL TRIAL: NCT04418219
Title: A Phase I/II Study of the SV-BR-1-GM Regimen in HLA Matched Metastatic Breast Cancer Patients in Combination With Pembrolizumab
Brief Title: Breast Cancer Vaccine in Combination With Pembrolizumab for Treatment of Persistent, Recurrent, or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding Discontinued
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20P.020; JT 14833 (Other: JeffTrial Number)
Record Dates: First submitted 2020-03-16; First posted 2020-06-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8; Recurrent Breast Carcinoma; Refractory Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; pembrolizumab; recombinant interferon alpha 2b-like protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SV-BR-1GM, pembrolizumab) (Experimental): Patients receive cyclophosphamide IV over 1-2 hours on day 1, SV-BR-1-GM ID on day 3, pembrolizumab IV over 30 minutes on day 5, and interferon-alpha-2b ID on days 5 and 7. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Biological: Allogeneic GM-CSF-secreting Breast Cancer Vaccine SV-BR-1-GM; Biological: Pembrolizumab; Biological: Recombinant Interferon Alpha 2b-like Protein; Other: Questionnaire Administration; Other: Quality of Life Assessment

INTERVENTIONS:
Drug: Cyclophosphamide — alkylating agent used in the treatment of several forms of cancer including leukemias, lymphomas and breast cancer.
Biological: Allogeneic GM-CSF-secreting Breast Cancer Vaccine SV-BR-1-GM — Breast Cancer Vaccine SV-BR-1-GM, Bria-IMT, GM-CSF Gene-transfected Breast Cancer Vaccine SV-BR-1-GM, SV-BR-1 Breast Cancer Cell Line Vaccine, SV-BR-1-GM, SV-BR-1-GM Vaccine
Biological: Pembrolizumab — 1374853-91-4, Immunoglobulin G4, Anti-(Human Programmed Cell Death 1); Humanized Mouse Monoclonal (228-L-proline(H10-S>P))gamma 4 Heavy Chain (134-218'')-disulfide with Humanized Mouse Monoclonal Kappa Light Chain Dimer (226-226'''':229-229'''')-bisdisulfide, Keytruda, Lambrolizumab, MK-3475, PEMBROLIZUMAB, SCH 900475
Biological: Recombinant Interferon Alpha 2b-like Protein — Novaferon, Recombinant IFN Alfa-2b-like Protein
Other: Questionnaire Administration — Ancillary studies
Other: Quality of Life Assessment — Ancillary studies

SUMMARY:
This phase I/II trial studies the side effects of a breast cancer vaccine (SV-BR-1-GM) and how well it works in combination with pembrolizumab for the treatment of breast cancer that is persistent, has come back (recurrent), or has spread to other places in the body (metastatic). Breast cancer vaccine SV-BR-1-GM is a human breast cancer cell line that has been genetically engineered to produce a substance called "GM-CSF" (granulocyte-macrophage colony stimulating factor) which occurs naturally in the body. GM-CSF is normally produced by white blood cells and helps the body develop immunity to disease-causing germs. Immunotherapy with monoclonal antibodies such as pembrolizumab may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Anti-cancer drugs such as cyclophosphamide may help boost the immune response. Interferon alpha 2b may help stimulate the immune system to fight cancer. This trial may help doctors see whether SV-BR-1-GM injections help boost the immune system and/or help control or help shrink breast cancer along with the other drugs that also boost the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of the allogeneic GM-CSF-secreting breast cancer vaccine SV-BR-1-GM (SV-BR-1-GM) regimen when administered in combination with pembrolizumab in patients with human leukocyte antigen (HLA) match. (Phase I) II. To evaluate the overall response rate of the SV-BR1-GM regimen in combination with pembrolizumab. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the non-progressive rate of the SV-BR-1-GM regimen in combination with pembrolizumab.

II. To evaluate the duration of response of the SV-BR-1-GM regimen in combination with pembrolizumab.

III. To evaluate immune responses elicited by the SV-BR-1-GM regimen when administered in combination with pembrolizumab.

IV. To evaluate patient and tumor characteristics that may be predictive of responses to the SV-BR-1-GM regimen when administered in combination with pembrolizumab.

V. To evaluate quality of life (QOL) in patients administered the SV-BR-1-GM regimen in combination with pembrolizumab by the Edmonton Symptom Assessment Survey.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) over 1-2 hours on day 1, SV-BR-1-GM intradermally (ID) on day 3, pembrolizumab IV over 30 minutes on day 5, and interferon-alpha-2b ID on days 5 and 7. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2-4 weeks and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have evidence of persistent, recurrent, or progressive metastatic breast cancer for which there is no known or established treatment available with curative intent, after failing at least two courses of community standard systemic treatment with chemotherapy (and endocrine therapy, if appropriate)

  * Human epidermal growth factor 2 (HER2) positive and estrogen receptor (ER) or progesterone receptor (PR) positive tumors: must be refractory to hormonal therapy (e.g., aromatase inhibitor, tamoxifen or fulvestrant) and previously treated with at least 1 regimen that includes at least two antiHER2 agents (e.g., trastuzumab and pertuzumab)
  * ER/PR positive, HER2 negative tumors: must be refractory to hormonal therapy (e.g. aromatase inhibitor, tamoxifen or fulvestrant) and previously treated with at least 2 chemotherapy containing regimens
  * HER2 positive and ER/PR negative tumors: must have failed at least 2 regimens including at least two anti-HER2 agents (e.g., trastuzumab and pertuzumab)
  * Triple negative tumors (defined as ER < 1%, PR < 1% as per American Society of Clinical Oncology College of American Pathologists [ASCO CAP] guidelines, HER2/neu 0-1 by immunohistochemistry [IHC] or negative by dual in situ hybridization [ISH]): Must have failed two other treatment lines including either a taxane and/or atezolizumab. Patients can have had atezolizumab (PD-L1 inhibitor) or PD-1 therapy previously
* Patients will only be eligible for this study if they have at least one human leukocyte antigen (HLA) match:

  * HLA-A*24:02
  * HLA-B*35:08
  * HLA-B*55:01
  * HLA-C*04:01
  * HLA-C*01:02
  * HLA-DRB3*01:01
  * HLA-DRB3*02:02
* Have expected survival of at least 4 months
* Have adequate performance status (Eastern Cooperative Oncology Group [ECOG] 0-1)
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) defined as spontaneous cessation of menstrual cycle for at least 12 months or surgical history of hysterectomy or bilateral salpingoopherectomy OR
  * A WOCBP who agrees to take appropriate precautions to avoid becoming pregnant during the treatment period and for at least 90 days plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* If any brain metastases, must have had prior radiation therapy for brain metastases
* Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology are allowed. The use of physiologic doses of corticosteroids may be approved after consultation with the principal investigator
* Absolute neutrophil count (ANC) >= 1500/uL (collected within 14 days prior to the start of study treatment)
* Platelets >= 100,000/uL (collected within 14 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (collected within 14 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 14 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase) [[SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase) [[SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (collected within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)

Exclusion Criteria:

* Concurrent or recent chemotherapy, radiotherapy, immunotherapy, or general anesthesia/major surgery within 4 weeks
* Patients must have recovered from all known or expected toxicities from previous treatment and passed a treatment-free "washout" period of 3 weeks before starting this program
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to enrollment
* Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline

  * Participants with =< grade 2 neuropathy and/or alopecia may be eligible
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g, FluMist) are live attenuated vaccines and are not allowed
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* History of clinical hypersensitivity to granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon-alpha-2b, yeast, beef, or to any components used in the preparation of SV-BR-1-GM
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Proteinuria >1+ on urinalysis or >1 gm/24hr
* Left ventricular ejection fraction (LVEF as determined by cardiac echo or multigated acquisition scan [MUGA] scan) below the normal limits of the institutions' specific testing range. This assessment may be repeated once at the discretion of the Investigator with the approval of the principal investigator
* New York Heart Association stage 3 or 4 cardiac disease
* A pleural or pericardial effusion of moderate severity or worse
* WOCBP who have a positive urine pregnancy test within 7 days prior to enrollment

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Women who are pregnant or nursing
* Patients with concurrent second malignancy. Persons with previous malignancies effectively treated and not requiring treatment for > 24 months are eligible, provided there is unambiguous documentation that current local recurrence or metastatic site represents recurrence of the primary breast malignancy
* Patients who are human immunodeficiency virus (HIV) positive (by self-report) or have clinical or laboratory features indicative of acquired immunodeficiency syndrome (AIDS)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] is detected) infection
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients who require systemic steroids at doses > 10 mg daily of prednisone or equivalent or any immunosuppressive drugs. Beta-blocker therapy, while not exclusionary, is discouraged and alternatives should be sought if possible. The beta-blocker might compromise use of epinephrine for the rare possibility of anaphylaxis
* Patients with a history of colitis
* Patients with severe psychiatric (e.g., schizophrenia, bipolar, or borderline personality disorder) or other clinically progressive major medical problems, unless approved by the principal investigator
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Patients may not be on a concurrent treatment clinical trial, unless approved by principal investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-21 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 1 year
  Toxicity will be determined using the Common Terminology Criteria for Adverse Events (CTCAE v 5.0).
Objective response rate (ORR) | up to 1 year
  Will be defined as complete response (CR), partial response (PR) or stable disease (SD) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-modified (i)RECIST. The method of Atkinson and Brown will be used to allow for the two-stage design.

SECONDARY OUTCOMES:
Non-progressive rate | Up to one year
  Defined as time to progression of disease, measured by CR, PR or SD per RECIST 1.1 and iRECIST. This will be estimated using the Kaplan-Meier method.
Durability of response | Up to one year
  Defined in time as time to progressive disease.
Delayed type hypersensitivity (DTH) skin tests | Up to 1 year
  Will be evaluated comparing pre-dose with post-dose samples using simple statistical testing (e.g. Student's t-Test).
T cell responses to SV-BR-1 | Up to 1 year
  Will be evaluated comparing pre-dose with post-dose samples using simple statistical testing (e.g. Student's t-Test).
Tumor expression of PD-L1 | Up to 1 year
Tumor expression of PD-L2 | Up to 1 year
Tumor expression of cancer/testis antigens such as PRAME | Up to 1 year
Type of breast cancer (estrogen receptor [ER] positive, HER2 positive, triple negative) | Up to 1 year
Edmonton Symptom Assessment Survey | Up to 1 year
  Assessment of nine symptoms commonly seen in cancer patients. Patients rate on scale of 0-10 with 0 meaning the symptom is absent and 10 meaning the worst possible severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States